CLINICAL TRIAL: NCT02340091
Title: A Randomized, Multi Center, Double-blind, Active-controlled, Matched Pairs Design Clinical Study to Evaluate the Efficacy and Safety of HA IDF Plus Versus HA IDF in Nasolabial Fold Injection
Brief Title: A Clinical Study to Evaluate the Efficacy and Safety of YVOIRE Classic Plus Versus YVOIRE Classic in Nasolabial Fold Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: LG-HACL012
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2015-01

CONDITIONS: Wrinkles
Keywords: facial nasolabial fold wrinkles

STUDY DESIGN:
Intervention Model Description: split-face design study. Subjects were decided by randomization which side of the face would be injected with the test device. According to this randomization result, the other side would be determined to be injected with a comparator. It was determined just by one randomization.
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- HA IDF plus (Experimental): cross-linked HA filler with lidocaine
  Interventions: Device: HA IDF plus
- HA IDF (Active Comparator): cross-linked HA filler without lidocaine
  Interventions: Device: HA IDF

INTERVENTIONS:
Device: HA IDF plus
  Arms: HA IDF plus
Device: HA IDF
  Arms: HA IDF

SUMMARY:
The objective of this study was to evaluate the efficacy and safety of HA IDF plus (with lidocaine) injected in the nasolabial fold compared to HA IDF (without lidocaine).

DETAILED DESCRIPTION:
The objective of this study was to confirm the superiority of HA IDF II plus (with lidocaine) injected in the nasolabial fold compared to HA IDF II (without lidocaine) in the improvement of local pain and evaluate the wrinkle-correcting effect, GAI and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged between 30 and 60
2. Those whose wrinkles in the treatment area (nasolabial fold) correspond to Stage 3 or 4 in the 5-stage Wrinkle Severity Rating Scale (WSRS) symmetrically
3. Those who were informed on the purpose, method, and effect etc. of this study and signed the informed consent form
4. Those who fell under any of the following 3 cases:

   1. Surgically sterile women
   2. Women in menopause over 2 years from the last menstruation, aged at least 45
   3. Among the women meeting neither of a nor b, those who agreed to use at least 2 contraception methods specified below (one of the barrier methods must be included) until 14 days after the last treatment with the investigational medical device

      * Barrier methods: Condom, diaphragm, cervical cap (pessary), spermicide
      * Hormonal methods: Pills, injection (depot), skin patch, hormonal implant (Implanon), vaginal ring
      * Intrauterine devices (IUDs): Cooper IUD (Loop), hormonal IUD (Mirena)
      * Natural methods: Basic body temperature, ovulation period, coitus interrupts, abstinent

Exclusion Criteria:

1. Those with a skin disease (skin infection, eczema, psoriasis, rosacea, herpes etc.) in the lower 2/3 part of the face in which the wrinkle evaluation may be affected
2. Patients who had been treated for a malignant tumor within 5 years prior to Visit 2 (randomization)*
3. Women in pregnancy or lactation
4. Those with the bilirubin level exceeding 1.5x of the upper limit of normal or the ALT/AST level exceeding 2.5x of the upper limit of normal
5. Those with the confirmed infection of syphilis or HIV
6. Those who had an anticoagulant therapy or antiplatelet therapy within 2 weeks prior to Visit 1 (screening)
7. Those who used a topical preparation (steroid, retinoid) in the facial area within 4 weeks prior to Visit 2 (randomization)
8. Those who experienced a deep chemical peeling or a laser procedure (including IPL) within 3 months prior to Visit 2 (randomization)
9. Those who experienced a non-permanent filler procedure or a cosmetic surgery in the face within 9 months prior to Visit 2 (randomization)
10. Those who had an implantation procedure with a permanent substance (silicone, PAAG, PMMA, CaHA etc.) in the treatment area (nasolabial fold )
11. Those currently with a streptococcal disease
12. Those with a history of severe allergy or hypersensitivity (anaphylaxis) judged as potentially affecting the clinical study
13. Those with a history of hypertrophic scar or keloid
14. Those with a history of bleeding disorder
15. Those with a hypersensitivity to the investigational medical device of this clinical study or lidocaine
16. Those who refused to agree not to use a local or systemic pain-relieving agent or other pain-relieving method (e.g.: ice pack) from the midnight of the treatment day with the investigational medical device through the post-measurement of the last VAS pain scale
17. Those who had participated in another clinical study within 1 month prior to Visit 1 (screening)
18. Those judged by the investigator as ineligible for this clinical study * Excluded were the patients with treated basal cell or squamous cell skin cancer or treated cervical cancer, of which the location is not the lower 2/3 part of the face.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2015-06 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 62 subject in total in 2 institutions period : Feb 2014~ May 2015
Pre-assignment Details: spilt-face design
  Subjects were decided by randomization which side of the face would be injected with the test device. According to this randomization result, the other side would be determined to be injected with a comparator. It was determined just by one randomization.
Groups:
- Subject Disposition: All Study Participants
Period: Overall Study
Arm/Group | Subject Disposition
Started | 62 (All Study Participants)
Completed | 60
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Demographic Charateristics: Subjects who were included in efficacy evaluation
Arm/Group | Demographic Charateristics
Number analyzed (Participants) | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.71 (7.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of the Subjects With at Least 10mm Difference in VAS Pain Scale Scores Within the Subject (VAS of the Control Medical Device - VAS of the Test Medical Device) Immediately After Treatment With the Investigational Medical Devices
Description: The degree of pain was evaluated by VAS (Visual Analog Scale), measuring the length from the left and to the mark by the subject in millimeter (mm) unit.
Time Frame: Visit 2 (week 0, immediately after treatment)
Measure: Number; unit: participants
Groups:
- Subjects With at Least a 10mm Difference in VAS: Subjects with at least a 10mm difference in VAS (HA IDF II - HA IDF II plus)
- Subjects With Below 10mm Difference in VAS: Subjects with below 10mm difference in VAS (HA IDF II - HA IDF II plus)
Arm/Group | Subjects With at Least a 10mm Difference in VAS | Subjects With Below 10mm Difference in VAS
Number analyzed (Participants) | 62 | 62
participants | 57 | 5
Statistical Analysis 1: Comparison: Subjects With at Least a 10mm Difference in VAS vs Subjects With Below 10mm Difference in VAS; Test type: Superiority; Subjects % with difference in VAS ≥ 10mm = 0.9194, 95% CI 2-sided [0.80 to 0.97]

ADVERSE EVENTS:
Time Frame: The Safety set consisted of the subjects who were treated with the investigational device at least once after Visit 2 (Randomization) and had a safety follow-up at least once
Description: The safety results were analyzed in the Safety set, and the safety was evaluated for the endpoints of local reactions, adverse events, vital signs and laboratory tests.
Groups:
- Safety: Subject who were injected with investigational medical device at least once.
  The 'Serious Adverse Events' and 'Other Adverse Events' described below occured in each subject regardless of the left or right of the injection site, and since all subjects were injected with both test device and comparator, it was not indicated which side the test device was injected.
Arm/Group | Safety
Serious Adverse Events (participants affected / at risk) | 1/62
Other Adverse Events (participants affected / at risk) | 5/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety (N=62)
nasopharyngitis (Infections and infestations) | 1 (1) — 'continuous' occurrence, the severity was 'Moderate', the relationship was 'Not related', and the outcome was 'Recovered'.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety (N=62)
Bronchitis (Infections and infestations) | 5 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other